CLINICAL TRIAL: NCT04389411
Title: Repurposing Montelukast for the Attenuation and Prophylaxis of Severe COVID-19 Symptoms: The COvid-19 Symptom MOntelukast (COSMO) Trial
Brief Title: The Covid-19 Outpatient Symptom Montelukast Oximetry Trial
Acronym: COSMO
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University (Other)
Collaborators: Segal Cancer Centre (Unknown); The McGill Practice Based Research Network (Unknown); Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Machelle Wilchesky, Assistant Professor, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 443807
Record Dates: First submitted 2020-05-13; First posted 2020-05-15 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Montelukast and placebo tablets will be over encapsulated before distribution to trial participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Montelukast (Experimental): 10mg Oral Montelukast once daily for 60 days
  Interventions: Drug: Montelukast 10mg
- Placebo (Placebo Comparator): Placebo.
  Interventions: Drug: Montelukast 10mg

INTERVENTIONS:
Drug: Montelukast 10mg — 10mg oral Montelukast will be taken daily for 60 days

SUMMARY:
Primary care physicians face limited availability of therapeutic options for the treatment of COVID-19 in the outpatient setting. Furthermore, monoclonal antibodies and antiviral therapies that are currently approved for use in the outpatient setting by Health Canada have excluded pregnant women and older adults from their clinical trials, are contraindicated for many patients, and most are prohibited for use by pregnant women. Identification of a safe, COVID-19 outpatient therapeutic with 20-year safety record remains urgently needed.

DETAILED DESCRIPTION:
Objectives: Our overarching objective is to determine the efficacy of oral montelukast versus placebo in reducing the duration and severity of COVID-19 symptoms among newly infected at-risk adults in the outpatient setting using a randomized controlled trial. Our two primary objectives are to compare the efficacy of oral montelukast versus placebo in reducing:

1. Symptom severity during the first 14 days of follow-up as measured by differences in mean FluPro PLUS scores and blood oxygen saturation SpO2 levels; and in reducing
2. C-Reactive Protein a biomarker of inflammation associated with severe COVID, obtained on days 3, 6, 9, and 14 of follow-up.

Our 7 secondary objectives of the COSMO Trial include evaluating the efficacy of Montelukast in improving: i) Duration of symptoms; ii) Interleukin IL-6; iii) Hypoxemia; iv) Symptom severity during the first 21 and 30 days of follow-up; and v) Healthcare services use in the 6 months post infection (including MD visits).

Hypothesis & Preliminary Evidence: We hypothesize that repurposing Montelukast to target suppression of NF- KappaB activation in COVID-19 positive patients will result in a corresponding reduction of Pro-inflammatory mediators, thereby attenuating cytokine production, and taming the cytokine storm, improved blood oxygen saturation, a reduction in hypoxia, mitigation of severe COVID-19 symptoms, and serve as a therapeutic for SARS-CoV-2 infections. Published articles authored by Dr. Geoff Tranmer (study PI) and others provide details of this hypothesis. A retrospective analysis of 92 COVID-19 hospitalized patients conducted by our study collaborators in the USA and Belgium provides evidence that patients who had received montelukast experienced significantly fewer events of clinical deterioration compared to patients not receiving montelukast (10% vs 32%, p= 0.022). More compelling, however, is the fact that montelukast is presently being used by a growing number of clinicians around the world on a compassionate basis for their patients and is currently the standard for COVID-19 patient care in some parts of the world.

Methods and Approaches: The COvid-19 Symptom Montelukast Outpatient (COSMO) Trial will be a parallel assignment, phase II, quadruple blinded, randomized, placebo-controlled trial of Montelukast for the treatment of SARS-CoV-2 infections. The study will include 250 recently infected pregnant or older adult outpatients at risk of severe disease who will be randomized to receive either treatment (20mg oral Montelukast) or matched placebo once daily, for 21 to 30 consecutive days. Patient symptoms will be monitored daily for a period of 30 days, after which follow-up will continue for an additional 60 days for outcomes such as duration of symptoms, resilience, functional status, quality of life. Healthcare services use will be evaluated at 6 months post enrollment. The study will be conducted at the Segal Cancer Center and at Quebec Primary Care Medicine Clinics with the utilization of the McGill Primary Care Practice Based Research Network and the Segal Cancer Centre clinical trials infrastructure, with recruitment directly within participating clinics.

Expertise and Support: We have developed a team that possesses extensive clinical and epidemiology experience. To date, we have gained support from our participating clinics, the PRBN, the CEO of a CIUSSS Network, clinical trial infrastructure (Segal Centre), and clinical trial support (IMS). We have also received have in-kind support from Masimo (Rad-5/5V hand-held stand-alone hospital grade Pulse Oximeters valued at $40,000 CAD to be used for 3x daily symptom reporting) and $5,000USD in cash support from an independent partner.

Outcomes: A therapeutic will remain necessary in the context of uncertain vaccine effectiveness, vaccine hesitancy and viral mutations. With positive results from the COSMO trial, we expect Montelukast to be recommended for COVID-19 outpatients given that it is safe, effective, and globally available

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed SARS-CoV-2 infection, defined as RT-PCR provincial laboratory confirmation;
2. Time from patient reported first symptoms date of enrollment <7 days;
3. Must be experiencing at least 1 COVID-19 symptom that is either continuing or increasing in severity
4. Severe disease risk factor requirements: i) Age 18-49: ≥3 risk factors ; ii) Age 50-59: ≥2 risk factors; iii) Age 60-69: ≥1 risk factor; iv) Pregnant or Age 70+: No requirements
5. Participants must agree to: i) Use assigned medication for a maximum of 60 days or until relief of symptoms; and ii) Complete the FLU-PRO PLUS and SpO2 daily diary and other study assessments during the course of follow-up.

Exclusion Criteria:

1. Any hospitalization for COVID-19 symptoms or complications prior to randomization;
2. Use of montelukast ≤ 30 days to screening;
3. Any contraindication to montelukast; and
4. Any condition (including the inability to swallow pills) which, in the opinion of the Principal Investigator, would prevent full participation in and compliance with the trial protocol, or would interfere with the evaluation of trial endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Symptom Severity | 14 days
  Symptom severity during the first 14 days of follow-up as measured by differences in mean FluPro PLUS scores
C-Reactive Protein | 14 days
  C-Reactive Protein a biomarker of inflammation associated with severe COVID, obtained on days 3, 6, 9, and 14 of follow-up

SECONDARY OUTCOMES:
Duration of symptoms | 90 days
  Duration of symptoms as measured by differences in mean FluPro PLUS scores
Interleukin IL-6 | 14 days
  Interleukin IL-6, a biomarker of inflammation associated with severe COVID, obtained on days 3, 6, 9, and 14 of follow-up
Hypoxemia incidence | 30 days
  Each participant will be provided with a Health Canada approved Masimo Rad 5/V pulse Oximeter upon enrollment. home pulse oximetry (SpO2) recorded 3 times daily for the first 30 days of follow-up. Hypoxemia will be defied as SpO2 <92% on room air for >5 minutes.
Hypoxemia | 30 days
  Differences in the means using the 2 lowest (validated) SpO2 values per patient
Functional Status | 30 days
  As measured using the Post-COVID-19 Functional Status Scale
Time to other serious COVID-19 complications | 12 weeks
  Complications will be defined as a composite endpoint including pneumonia, ARDS sepsis/septic shock, cardiomyopathy or arrhythmia, acute kidney injury, and secondary bacterial infections.
Hospitalization | 6 months
  Hospital visits- (healthcare services use component)
Medications | 6 months
  Medication use- (healthcare services use component)
Physician Visits | 6 months
  Visits to primary care and specialists- (healthcare services use component)
Cost-Effectiveness | 6 months
  Comparison of healthcare services use costs

CONTACTS AND LOCATIONS:
Overall Officials: Machelle Wilchesky, PhD, Principal Investigator — Lady Davis Institute and McGill University; Geoffrey Tranmer, PhD, Principal Investigator — University of Manitoba; Roland Grad, MDCM MSc FCFP, Principal Investigator — Herzl Family Practice Centre and McGill University

IPD SHARING:
Plan to Share IPD: Yes
COSMO Trial Data Governance Plan: We have designed the COSMO Trial to uphold the FAIR principles such that the research data derived will be Findable, Accessible, Interoperable, and Reusable. The raw data from this study, once removed of identifiers, will be posted to a public data sharing resource to allow the data to be used and understood by the wider scientific community. The precise platforms and open access data repositories will be determined once the data is ready, but candidate platforms include github and the Google COVID-19 data sharing platform.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: We will make this data available within 12 months of completion of data collection.
Access Criteria: Undetermined.

REFERENCES:
- [Background] Sanghai N, Tranmer GK. Taming the cytokine storm: repurposing montelukast for the attenuation and prophylaxis of severe COVID-19 symptoms. Drug Discov Today. 2020 Dec;25(12):2076-2079. doi: 10.1016/j.drudis.2020.09.013. Epub 2020 Sep 16. PMID 32949526